CLINICAL TRIAL: NCT03753295
Title: The Effect of BMI on Hand Grip Force in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Wafaa Mahmoud Amin (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Wafaa Mahmoud Amin, Lecturer, University of Jazan
Organization: University of Jazan (Other Government)
Other Study IDs: 27704112500
Record Dates: First submitted 2018-11-23; First posted 2018-11-26 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Motor Activity; Overweight and Obesity; Hand Injuries
Keywords: BMI, Hand Grip, Healthy Adults
MeSH Terms: conditions — Motor Activity; Overweight; Obesity; Hand Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I (normal subjects): 30 individuals (15 male, and 15 female students) with (BMI<25 kg/m2). Hand grip force will measured using Baseline Hydraulic Hand Dynamometer.
  Interventions: Diagnostic Test: Hand Grip Force
- Group II (overweight subjects): 30 individuals (15 male, and 15 female students) with (BMI, 25-30 kg/m2). Hand grip force will measured using Baseline Hydraulic Hand Dynamometer.
  Interventions: Diagnostic Test: Hand Grip Force
- Group III (obese subjects): 30 individuals (15 male, and 15 female students) (BMI>30 kg/m2). Hand grip force will measured using Baseline Hydraulic Hand Dynamometer.
  Interventions: Diagnostic Test: Hand Grip Force

INTERVENTIONS:
Diagnostic Test: Hand Grip Force — For measuring the grip strength, the subjects will be asked to sit on a chair with their hip joint flexed at 90 degree, and shoulder joint in a neutral position.
  The elbow is fixed at 90 degree flexion, forearm in a neutral position, and wrist at 0 to 15 degree radial deviation.
  The test will be performed twice, and the higher value between the two measurements will be selected.
  The subjects will be allowed a rest time of more than 5 minutes after the first measurement to avoid examiner bias and to decrease physical stress

SUMMARY:
This study will be conducted to investigate the effect of BMI on hand grip force in healthy subjects. The participants in this study will be 90 healthy subjects with right dominant lower limb (49 females and 49 males) they will be recruited from College of Applied Medical Sciences, Jazan University.

DETAILED DESCRIPTION:
Subjects will be categorized according to BMI into three groups:

Group I (normal subjects): 30 individuals (15 male, and 15 female students) with (BMI<25 kg/m2) Group II (overweight subjects): 30 individuals (15 male, and 15 female students) with (BMI, 25-30 kg/m2).

Group III (obese subjects): 30 individuals (15 male, and 15 female students) (BMI>30 kg/m2).

Baseline hydraulic hand dynamometer: (Fabrication Enterprises Incorporated, White Plains,New York, USA) will be used to measure the hand grip strength and pinch strength

ELIGIBILITY:
Inclusion Criteria:

1. Subjects would not have any diseases of the central nervous system.
2. Subjects would not have any orthopedic disorders either of the trunk or the lower limbs in the previous year.
3. None of the subjects has history of balance training ( Erkmen et al., 2010, Li Li, 2012) .

Exclusion Criteria:

1. Sign of foot pain, reduced tactile and thermal foot sensibility.
2. Peripheral neuropathy.
3. A history of previous back or abdominal surgery/injury
4. A history of patellofemoral pain syndrome, plantar fasciitis, and back pain .
5. Limb-length discrepancy, and anterior or posterior tibialis dysfunction.
6. Evidence of a systemic or musculoskeletal disease within the past six months (AlAbdulwahab & Kachanathu, 2016).

Ages: 19 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: 90 healthy male and female students with age 19 to 25 years old, and right dominant hand, will be recruited from the College of Applied Medical Sciences, Jazan University.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Hand Grip Force of the Right Dominant Hand in The Three Groups | 10 minutes
  Hand Grip strength will be measured in three groups and comparison between them will be made
Comparison of Hand Grip Force between Both Arms in three Groups | 20 minutes
  Measurement of both right dominant hand and left hand will be measured in the three groups and compared with each other.

SECONDARY OUTCOMES:
the effect of gender on the hand grip | 10 minutes
  measurement of hand grip force of the right dominant hand will be taken for both male and females in the three subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Riyadh, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided